CLINICAL TRIAL: NCT02179294
Title: A Randomised Controlled Trial of Remifentanil Intravenous Patient Controlled Analgesia (PCA) Versus Intramuscular Pethidine for Pain Relief in Labour
Acronym: RESPITE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Heartlands Hospital (Unknown); Good Hope Hospital (Unknown); Birmingham Women's NHS Foundation Trust (Other Government); York Hospital (Unknown); University Hospital of North Midlands (Unknown); Frimley Park Hospital (Unknown); Bradford Royal Infirmary (Other); Stoke Mandeville Hospital (Unknown); Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other); Medway Maritime Hospital (Unknown); Northwick Park Hospital (Other); Homerton University Hospital (Unknown); City Hospital Birmingham (Unknown); Warwick Hospital (Unknown); University Hospital Coventry (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_12-151; 2012-005257-22 (EudraCT Number)
Record Dates: First submitted 2014-06-11; First posted 2014-07-01 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Pain Relief in Labour
Keywords: Pain relief; Labour; Child birth; Anaesthetics
MeSH Terms: interventions — Meperidine; Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pethidine (Active Comparator): Pethidine is pain relief in labour
  Interventions: Drug: Pethidine
- Remifentanil (Active Comparator): Remifentanil intravenous patient controlled analgesia
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Pethidine — 100mg by intramuscular injection, up to 4 hourly in frequency (up to a maximum of 4 doses). The maximum dose being 400mg in 24 hours.
  Other Names: Meperidine
  Arms: Pethidine
Drug: Remifentanil — Dedicated intravenous cannula for remifentanil administration PCA protocol
  * PCA bolus remifentanil 40 μg
  * Lockout interval 2 minutes
  In the event of excess sedation being recorded by regular observation of respiratory function, the regimen will be altered by reduction of the remifentanil bolus dose to 30 μg with a lock-out interval of 2 minutes.
  Other Names: Ultiva
  Arms: Remifentanil

SUMMARY:
Childbirth can be an extremely painful and the provision of pain relief during labour is a vital component of a positive maternal experience. The majority of women who deliver in modern obstetric units choose a pharmacological method of pain relief, including Entonox, the injection of opioids or epidural placement. The commonest opioid used in labour is pethidine administered by intramuscular (im) injection. The effectiveness of pain relief provided by pethidine has long been challenged. Its shortcomings are more serious when set against known side effects including maternal sedation, nausea and potential transfer across the placenta to the foetus. More than a third of women who receive pethidine subsequently require an epidural due to inadequate pain relief. Epidurals provide highly effective pain relief, but increase the risk of a forceps or suction delivery resulting in prolonged hospital stay. Therefore, there is a clear need for a safe, effective, easy to administer analgesic alternative.

DETAILED DESCRIPTION:
Patient Controlled Analgesia (PCA) comprises drug administration into an intravenous drip with a small dose given each time a woman presses a button, giving her control over her own pain relief. The pump is programmed to ensure that the maximum dose allowable is within the safe range. This form of delivery of pain relief matches the drug dose to pain sensation within the relevant time frame, which is not possible using a single dose intramuscular injection. Whilst PCA is in widespread use for acute pain relief it has only a limited role in obstetrics. The most common drug given by PCA is morphine, however, since it has a long duration of action and crosses the placenta, the potential for accumulation in the foetus and consequent neonatal sedation at delivery restricts its utility (within obstetrics) to contexts where neonatal status is not relevant, such as intra-uterine foetal death or foetal abnormality incompatible with survival.

Remifentanil is a novel synthetic opioid with a very rapid onset (blood-brain equilibration 1.2-1.4 minutes) and short duration of action (context specific half-life 3 minutes), giving it an analgesic profile which potentially makes it ideal for providing pain relief over 1-2 uterine contractions after a single intravenous dose. It is subject to rapid redistribution and metabolism by non-specific blood and tissue esterases negating the potential for accumulation in mother or foetus. Administration of remifentanil by PCA has been investigated in several small studies in comparison to pethidine and shown to provide useful, although not complete, pain relief in labour.10-12 Thus far, there is no evidence of detrimental neonatal effects in comparison to other opioids.

ELIGIBILITY:
Inclusion Criteria:

Women who are admitted to labour ward who fulfil all the following criteria will be eligible to be randomised:

* Requesting systemic opioid analgesia
* 16 years of age or older
* Beyond 37 weeks gestation
* In established labour, defined as regular painful contractions, irrespective of cervical dilatation, with vaginal birth intended
* Able to understand all information (written and oral) presented (using an interpreter if necessary)
* Not participating in any other clinical trial of a medicinal product
* Live, singleton pregnancy with cephalic presentation

Exclusion Criteria:

* Contraindication to epidural analgesia
* Contraindication to intramuscular injection
* History of a previous adverse reaction to pethidine or remifentanil
* Patients taking long term opioid therapy including Methadone
* Systemic pain relief opioid in the last 4 hours administered by intravenous or intramuscular injection. (Oral medications comprising opioids alone or in combination preparations, administered in this 4 hour period, are permitted).

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2014-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The proportion of women who receive epidural analgesia for pain relief in labour, in each group, after randomisation. | At labour
  The proportion of women who receive epidural analgesia for pain relief in labour, in each group, after randomization.

SECONDARY OUTCOMES:
• The effectiveness of pain relief provided by each technique, quantified by Visual Analogue Scale | Post natally - Average of 2-3days after delivery
  • The effectiveness of pain relief provided by each technique, quantified by Visual Analogue Scale
The incidence of maternal side effects | Post Natally - Average of 2-3days after delivery
  The incidence of maternal side effects including
  * Excessive sedation score
  * Oxygen Saturation <94% whilst breathing room air
  * Nausea requiring anti-emetic administration
  * Requirement and indication for supplemental oxygen
  * Respiratory Depression (Respiratory rate < 8 breaths/minute)
Delivery mode (Spontaneous, Instrumental Vaginal, Caesarean Section) | Post Natally - Average of 2-3days after delivery
  Delivery mode (Spontaneous, Instrumental Vaginal, Caesarean Section)
Incidence of foetal distress requiring delivery | Post Natally - Average of 2-3days after delivery
  Incidence of foetal distress requiring delivery
Neonatal status at delivery | Post Natally - Average of 2-3days after delivery
  Neonatal status at delivery:
  * Apgar score at 5 minutes
  * Incidence of foetal acidosis determined by umbilical cord gas analysis
  * Requirement for neonatal resuscitation
  * Incidence of and indication for admission to neonatal care
Rate of initiation of breast feeding within the first hour of birth | Post Natally - 1 hour after delivery
  Rate of initiation of breast feeding within the first hour of birth
Maternal satisfaction with childbirth experience determined by postpartum questionnaire prior to discharge from the delivery ward | Post Natally - Average of 2-3days after delivery
  Maternal satisfaction with childbirth experience determined by postpartum questionnaire prior to discharge from the delivery ward
Maternal birth experience determined by qualitative telephone interview up to six weeks postpartum | Up to 6 weeks post-partum
  Explore and compare women's birth experiences up to six weeks postpartum via qualitative telephone interview (Post-Natal sub-study)
Maternal perceptions of pain relief determined by qualitative telephone interview up to six weeks postpartum | Up to 6 weeks post-partum
  Explore and compare women's perceptions of pain relief up to six weeks postpartum via qualitative telephone interview (Post-Natal sub-study)
Infant feeding behaviours determined by qualitative telephone interview up to six weeks postpartum | Up to 6 weeks post-partum
  Explore and compare infant feeding behaviours up to six weeks postpartum via qualitative telephone interview (Post-Natal sub-study)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew JA Wilson, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Birmingham Clinical Trials Unit, Birmingham, West Midlands, United Kingdom

REFERENCES:
- See also: Trial website — http://www.birmingham.ac.uk/respite